CLINICAL TRIAL: NCT05191706
Title: A Phase 3/4, Prospective, Randomized, Active Treatment-Controlled, Parallel-Design, Multicenter Study to Evaluate the Safety of DEXYCU for the Treatment of Inflammation Following Ocular Surgery for Childhood Cataract
Brief Title: Evaluate the Safety of DEXYCU for the Treatment of Inflammation Following Ocular Surgery for Childhood Cataract
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: EyePoint Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EYP-DIP-001
Record Dates: First submitted 2021-12-13; First posted 2022-01-13 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Cataract
Keywords: pediatric; cataract
MeSH Terms: conditions — Cataract | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Active Treatment-Controlled, Parallel-Design, Multicenter Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- DEXYCU (dexamethasoneintraocular suspension) 9% (Experimental): A single 0.005-mL anterior chamber injection of DEXYCU (dexamethasoneintraocular suspension) 9%, equivalent to 517mcg dexamethasone.
  Interventions: Drug: Dexamethasone
- Prednisolone acetate ophthalmic suspension (USP) 1% (Active Comparator): Active treatment control, prednisolone acetate ophthalmic suspension (USP) 1%, four times daily (QID) for 28days, followed by a treatment taper at the investigator's discretion.
  Interventions: Drug: Prednisolone Acetate Ophthalmic

INTERVENTIONS:
Drug: Dexamethasone — single anterior chamber injection
  Arms: DEXYCU (dexamethasoneintraocular suspension) 9%
Drug: Prednisolone Acetate Ophthalmic — topical administration four times a day for 28 days, followed by treatment taper
  Arms: Prednisolone acetate ophthalmic suspension (USP) 1%

SUMMARY:
A Phase 3/4, Prospective, Randomized, Active Treatment-Controlled, Parallel-Design, Multicenter Study to Evaluate the Safety of DEXYCUfor the Treatment of Inflammation Following Ocular Surgery for Childhood Cataract

ELIGIBILITY:
Inclusion Criteria:

* Undergoing uncomplicated cataract surgery with or without a posterior chamber intraocular lens (IOL) implantation.
* If a contact lens is used for correction of post-operative aphakia, it must be a silicone elastomer lens or a rigid gas permeable lens (no water content).
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Presence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, endocrine, neurological, psychiatric, respiratory, or other medical condition that could increase the risk to the subject as determined by the investigator.
* Has a post-traumatic cataract.
* Presence of active or suspected viral, bacterial, or fungal disease in the study eye.
* Ocular hypertension with an IOP in the study eye >25 mmHg at Screening with or without treatment with anti-glaucoma monotherapy.
* Subjects who have received a periocular corticosteroid injection in the study eye in the 3 months prior to Screening.
* Subjects who have received any intravitreal corticosteroid delivery vehicle (eg, Retisert®, Ozurdex®, Iluvien®) in the study eye at any time.
* Other protocol-specified exclusion criteria may apply

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Grade of anterior chamber cells (ACC) | Post-Operative Day 14

SECONDARY OUTCOMES:
Grade of anterior chamber flare (ACF) | Post-Operative Day 14

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - EyePoint Investigational Site, Huntington Beach, California
  - EyePoint Investigational Site, Palo Alto, California
  - EyePoint Investigative Site, Boston, Massachusetts
  - EyePoint Investigational Site, Jackson, Mississippi
  - EyePoint Investigational Site, Omaha, Nebraska
  - EyePoint Investigational Site, Buffalo, New York
  - EyePoint Investigative Site, New York, New York
  - EyePoint Investigational Site, Rochester, New York
  - EyePoint Investigational Site, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No